CLINICAL TRIAL: NCT03079349
Title: Randomized Controlled Study of a Remote Flipped Classroom Neuro-Otology Curriculum
Brief Title: Online Distance Learning Outcomes Compared to Traditional Classroom Learning in Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CI #20170222001
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Educational Problems
MeSH Terms: interventions — Early Medical Intervention

STUDY DESIGN:
Intervention Model Description: Subjects were randomized into a "control" group attending a traditional classroom and a "trial" group of equal numbers participating in an online synchronous Internet streaming classroom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Classroom (Active Comparator): Medical Education
  Interventions: Other: Medical Education; Other: Medical Intervention
- Online Synchronous Classroom (Experimental): Medical Education
  Interventions: Other: Medical Education; Other: Medical Intervention

INTERVENTIONS:
Other: Medical Education — All candidates in the Active Comparator: Traditional Classroom will take a pre course test of the subject material followed by two 9-hour and one 8-hour educational sessions given over 3 consecutive days. Following the educational sessions all candidates in the Active Comparator: Traditional Classroom will take a post course test.
Other: Medical Intervention — All candidates in the Experimental: Online Synchronous Classroom will take a pre course test of the subject material followed by two 9-hour and one 8-hour educational sessions given over 3 consecutive days. Following the educational sessions all candidates in theExperimental: Online Synchronous Classroom will take a post course test.

SUMMARY:
To test whether the investigator's educational methodology is associated with increasing learning of participants. The investigators second objective is to test the hypothesis that learning in an online classroom would result in similar outcomes as the traditional classroom.

DETAILED DESCRIPTION:
Subjects will be randomized into a "control" group attending a traditional classroom and a "trial" group of equal numbers participating in an online synchronous Internet streaming classroom.

Main outcome measures: Pre and post multiple choice examinations of Vestibulo-Ocular Reflex (VOR), Movement, Head Turns, Head Tremor, Neurodegeneration, Inferior Olivary Complex, Collateral Projections, Eye Movement Training, Visual Saccades, Head Saccades, Visual Impairment, Walking Speed, Neuroprotection, Autophagy, Hyperkinetic Movement, Eye and Head Stability, Oscilllatory Head Movements, Gaze Stability, Leaky Neural Integrator, Cervical Dystonia, Interstitial Nucleus of Cajal (INC) and Head Tilts, Visual Pursuits, Optokinetic Stimulation, Vestibular Rehabilitation.

Methods: All candidates will take a pretest examination of the subject material. Two 9-hour and one 8-hour sessions over 3 consecutive days will be given live in the classroom or synchronously in the online classroom using the Adobe Connect e-learning platform. Subjects randomized to the online classroom will attend the lectures in a location of their choice and will view the sessions live on the Internet. A posttest examination will be given to all candidates after completion of the course.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Health Care Professional, Active Practice

Exclusion Criteria:

* Non Licensed Health Care Professional, Non Active Practice

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Pretest and Posttest scores | 3 days
  Pre course test scores compared to Post course test scores

SECONDARY OUTCOMES:
Traditional vs Online Classroom Learning Scores | 3 days
  Pre course learning scores compared to Post course learning scores compared for traditional classroom and synchronous online learning classroom

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Bedfordshire Centre for Mental Health Research in Association with the University of Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrick FR, Abdulrahman M, Hankir A, Zayaruzny M, Najem K, Lungchukiet P, Edwards RA. Randomized Controlled Study of a Remote Flipped Classroom Neuro-otology Curriculum. Front Neurol. 2017 Jul 24;8:349. doi: 10.3389/fneur.2017.00349. eCollection 2017. PMID 28790966